CLINICAL TRIAL: NCT02845154
Title: Intermittent Anti-grade Portal and Graft Purge Ameliorates Post-reperfusion Syndrome in Living Donor Liver Transplantation Recipients. A Prospective, Randomised Controlled Trial
Brief Title: Intermittent Portal and Graft Purge in Living Donor Liver Transplantation
Acronym: IPLDLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, Professor of Anesthesia and Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDLDPURGE
Record Dates: First submitted 2015-10-16; First posted 2016-07-27 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2016-12

CONDITIONS: Hypotension; Ischemia Reperfusion Injury
Keywords: Ischemia reperfusion; post-reperfusion syndrome; living donor liver transplantation; patient outcome
MeSH Terms: conditions — Hypotension; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (bolus purge) (Active Comparator): The portal vein clamp will be totally released after end of portal vein anastomosis and all graft and portal blood contents are allowed free and complete access to the systemic circulation via the inferior vena cave
  Interventions: Other: bolus purge
- Intermittent Purge (Experimental): The portal clamp will be released in situ for 5 seconds to allow purge of the graft and portal contents into the systemic circulation, followed by 30 seconds of portal clamping again. This will be followed by another two cycles of 5 seconds declamping and 30 seconds clamping , then, the portal clamp will be completely released.
  Interventions: Other: Intermittent purge

INTERVENTIONS:
Other: bolus purge — complete and uninterrupted purge
  Arms: Control (bolus purge)
Other: Intermittent purge — intermittent portal purge
  Arms: Intermittent Purge

SUMMARY:
Post-reperfusion syndrome and ischemia-reperfusion insult are a common well-known complication in liver transplantation. Several trials investigated variables that my contribute to the generation of these two complications for reducing their incidence and magnitude. The investigators will investigate the effect of acute conditioning of the recipients circulation to the vasoactive mediators in the graft as well as the congested intestine through intermittent purging of graft contents into the patient's systemic circulation in living donor liver transplantation.

DETAILED DESCRIPTION:
Patients are subjected to living donor liver transplantation. In this type of grafts, cold ischemia time is minimal and the graft contents of preservative solution are less than cadaveric grafts. The investigators in the current research use HTC as a preservative solution. These factors justified the possibility of purging the graft and portal blood contents into the patient systemic circulation. The exposure to these fluids in this trial will be in an intermittent manner: the portal vein will be declamped for 5 seconds followed by 30 seconds of portal clamping. This will be repeated twice. The primary outcome objective in this trial will be the incidence of post-reperfusion syndrome. Secondary objectives include the severity of PRS, the incidence and severity of ischemia-reperfusion injury, graft and patient's survival.

ELIGIBILITY:
Inclusion Criteria:

* living donor liver transplantation recipients

Exclusion Criteria:

* Non

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Post-reperfusion syndrome | 5 minutes after portal declamping
  Reduced Mean arterial blood pressure to the predefined value

SECONDARY OUTCOMES:
Graft ischemia reperfusion injury | one week post-operative
  Pathological assessment of IR injury based on Suzuli score
Severity of post-reperfusion syndrome | 5 minutes after portal declamping
  % decrease in Mean arterial blood pressure
One month patient mortality | one month post-operative
  Mortality within one post-operative month

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, MD, Study Director — Mansoura Faculty of Medicine
Locations (3):
- Egypt (3):
  - Liver transplantation program - Gastroenterology surgical center, Al Mansurah, Dakahlia Governorate
  - Liver transplantation project - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate
  - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No